CLINICAL TRIAL: NCT01395901
Title: A Multicenter, Double-blind, Double-dummy, Randomized, Parallel Group, Stratified Study to Evaluate the Efficacy and Safety of a Single IV Dose of Palonosetron Compared to a Single IV Dose of Ondansetron to Prevent Postoperative Nausea and Vomiting in Pediatric Patients.
Brief Title: Safety and Efficacy of Palonosetron IV to Prevent Postoperative Nausea and Vomiting in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PALO-10-14
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Results first posted 2014-07-30 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2014-07

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Prevention of Postoperative Nausea and Vomiting; Palonosetron; Ondansetron; Pediatric
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting | interventions — Palonosetron; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palonosetron and placebo to Ondansetron (Experimental): Intervention: Drug: Palonosetron
  Interventions: Drug: Palonosetron; Drug: Placebo to Ondansetron
- Ondansetron and placebo to Palonosetron (Active Comparator): Intervention: Drug: Comparator: Ondansetron
  Interventions: Drug: Ondansetron; Drug: Placebo to Palonosetron

INTERVENTIONS:
Drug: Palonosetron — Single dose Palonosetron IV 1 mcg/kg (up to a maximum total dose of 0.075 mg)
  Arms: Palonosetron and placebo to Ondansetron
Drug: Ondansetron — Single dose Ondansetron IV:
  * 0 months to 12 years dose: 0.1 mg/kg for ≤ 40 kg and 4 mg for >40 kg;
  * 13 years to less than 17 years dose: 4 mg
  Arms: Ondansetron and placebo to Palonosetron
Drug: Placebo to Ondansetron
  Arms: Palonosetron and placebo to Ondansetron
Drug: Placebo to Palonosetron
  Arms: Ondansetron and placebo to Palonosetron

SUMMARY:
The primary objective of this study is to evaluate the efficacy of a single palonosetron IV dose compared to a single ondansetron IV dose in the prevention of postoperative nausea and vomiting through 24 hours after surgery in children aged from neonates up to less than 17 years undergoing elective surgical procedures requiring general intravenous anesthesia. The secondary objective is to evaluate the safety and tolerability of IV palonosetron in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged from full term neonate to less than 17 years.
* In-patient or out-patient scheduled to undergo one of the following procedures:

  * ear, nose and throat surgery (e.g., tonsillectomy, adenoidectomy, myringotomy),
  * eye surgery (e.g. strabismus, vitreoretinal, cataract surgery),
  * urological surgery (e.g. orchidopexy, varicocoele),
  * plastic reconstructive surgery (e.g. cleft lip/cleft palate, burn procedures involving the scalp),
  * hernia repair,
  * orthopedic surgery (e.g. foot and ankle deformities, arthroscopic surgeries, ACL surgery),.
  * cardiac surgery,
  * neurosurgery.
* Patient is scheduled to undergo surgery requiring general intravenous anesthesia
* Patient is scheduled to receive nitrous oxide during the maintenance phase of anesthesia
* Patient weighs at least 3.2 kg
* ASA physical status I, II or III
* Fertile patients (male or female) must use reliable contraceptive measures
* Female patients who have attained menarche must have a negative pregnancy test at the screening visit (Visit 1) and at study treatment visit (Visit 2)
* For patients with known hepatic impairment: in the Investigator's opinion, the impairment does not jeopardize the patient's safety during the study
* For patients with known renal impairment: in the Investigator's opinion, the impairment does not jeopardize the patient's safety during the study

Exclusion Criteria:

* Lactating females
* Patient aged ≤6 years who received any investigational drug within 90 days prior to Day 1, or patient aged >6 years who received any investigational drug within 30 days prior to Day 1 or is expected to receive investigational drugs prior to study completion.
* Patient having participated in any previous trial with palonosetron.
* History of allergy to any components or any other contraindications to the use of any 5-HT3 receptor antagonists
* Patient to undergo emergency surgery
* Patient scheduled to receive regional anesthesia (lumbar, epidural, spinal) alone or in conjunction with general intravenous anesthesia
* Patient scheduled to receive laryngeal mask anesthesia
* Patient scheduled to receive propofol during the maintenance phase of anesthesia
* Patient suffering from any concomitant disease uncontrolled by therapy, which, in the judgment of the Investigator, could compromise the outcome of surgery
* Patient with history of gastro-esophageal reflux (except for patients up to 12 months)
* Patient with ongoing vomiting from any organic cause
* Patient having experienced any vomiting, retching, or nausea within 24 hours prior to the administration of the study drug

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 670 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (12):
  - Shoals Clinical Research Associates, Florence, Alabama
  - Shoals Medical Research, LLC, Sheffield, Alabama
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Bascom Palmer Eye Institute - University of Miami, Miami, Florida
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - CRC of Jackson, Jackson, Mississippi
  - Cooper University Hospital, Camden, New Jersey
  - The University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Clinical Trial Developers, Cincinnati, Ohio
  - Texas Orthopedic Specialist, P.A, Grapevine, Texas
  - Memorial Hermann Hospital, Houston, Texas
- Argentina (2):
  - CEMIC, Otorhinolaryngology Department, Buenos Aires
  - Istituto Medico Rio Cuarto, Río Cuarto
- Czechia (6):
  - University Hospital Brno - Children's Medical Centre, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - University Hospital Pilsen- Paediatric Clinic, Plzen-Lochotin
  - University Hospital Motol, Prague
  - Hospital Znojmo, State-Funded Organisation, Department of Pediatrics, Znojmo
- Hungary (5):
  - Semmeleis University, Budapest
  - St Istvan and St Laszlo Corporate Hospital; Paediatric Intensive Care Unit, Budapest
  - The Municipal Council's St Janos Hospital and North Buda United Hospitals; Central Anaesthesiology and Intensive Care Unit, Budapest
  - St Panthaleon Hospital; Central Department of Anaesthesiology and Intensive Care Unit, Dunaújváros
  - Pandy Kalman County Hospital; Department of Central Anaesthesiology and Intensive Care Unit, Gyula
- Poland (5):
  - Department of Pediatric Surgery and Urology of Medical University of Gdansk, Gdansk
  - Department of Pediatric Anesthesiology and Intensive Care, Lodz
  - Department of Pediatric Anesthesiology and Intensive Care, Lublin
  - Department of Intensive Care and Anesthesiology, Olsztyn
  - Department of Pediatric Surgery, Wroclaw
- University Pediatric Hospital, San Juan, Puerto Rico
- Russia (5):
  - State Healthcare Institution Arkhangelsk Regional Children's Hospital, Arkhangelsk
  - Federal State Institution: St. Petersburg Research Institute of Ear, Throat, Nose and Speech under the MoH Care and Social Development of the Russian Federation, Saint Petersburg
  - International Clinic MEDEM, Saint Petersburg
  - St. Petersburg State Pediatric Medical Academy, Saint Petersburg
  - Yaroslavl Region State Healthcare Institution, Yaroslavl
- Ukraine (8):
  - Dnipropetrovsk Regional Childrens Clinical Hospital, Dnipropetrovsk
  - Regional Childrens Clinical Hospital, Donetsk
  - Ivano-Frankivsk Regional Childrens Clinical Hospital, Ivano-Frankivsk
  - City Clinical Hospital n#30, Kharkiv
  - Research and Development Center for Prophylactic and Clinical Medicine, Kyiv
  - National Specialized Childrens Hospital OKHMATDYT, Kyiv
  - V.P. Filatov Institute of Eye Diseases and Tissue Therapy, Odesa
  - Zaporizhia Regional Clinical Childrens Hospital, Zaporizhia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 44 sites were initiated in seven countries with 12, 9, 5, 5, 5, 6 and 2 investigative sites in the United States, Ukraine, Hungary, Poland, Russia, Czech Republic and Argentina. Patients were enrolled into the study by 39 out of 44 Investigators enrolling at least one patient.
Groups:
- Palonosetron and Placebo to Ondansetron: Intervention: Drug: Palonosetron
  Palonosetron: Single dose Palonosetron IV 1 mcg/kg (up to a maximum total dose of 0.075 mg)
  Placebo to Ondansetron
- Ondansetron and Placebo to Palonosetron: Intervention: Drug: Comparator: Ondansetron
  Ondansetron: Single dose Ondansetron IV:
  * 0 months to 12 years dose: 0.1 mg/kg for ≤ 40 kg and 4 mg for >40 kg;
  * 13 years to less than 17 years dose: 4 mg
  Placebo to Palonosetron
Period: Overall Study
Arm/Group | Palonosetron and Placebo to Ondansetron | Ondansetron and Placebo to Palonosetron
Started | 336 (Randomized Population) | 334 (Randomized Population)
Completed | 326 (Treated patients completing the study) | 329 (Treated patients completing the study)
Not Completed | 10 | 5
Not completed — Lost to Follow-up | 4 | 0
Not completed — Randomized but not received study drug | 5 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal of consent | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Palonosetron and Placebo to Ondansetron | Ondansetron and Placebo to Palonosetron | Total
Number analyzed (Participants) | 331 | 330 | 661
Age, Customized [Number; unit: participants]
  <2 years | 22 | 24 | 46
  2 <6 years | 124 | 123 | 247
  6 <12 years | 117 | 117 | 234
  12 <17 years | 68 | 66 | 134
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 129 | 261
  Male | 199 | 201 | 400
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 21 | 45
  Not Hispanic or Latino | 307 | 309 | 616
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 12 | 25
  White | 315 | 312 | 627
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Complete Response
Description: Complete Response was defined as no vomiting, no retching, and no use of antiemetic rescue medication during the first 24 hours postoperatively, starting at T0. Time 0 (T0) was defined as the time when the patient wakes up and is able to show any active reaction postoperatively.
Time Frame: 0-24 hours after T0
Population: The Full Analysis Set (FAS) included all randomized patients who received the active study drug, general anesthesia and surgery (evaluable patients). Following the intent-to-treat principle, patients were assigned to the study treatment arm according to their randomized treatment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Palonosetron and Placebo to Ondansetron | Ondansetron and Placebo to Palonosetron
Number analyzed (Participants) | 331 | 330
percentage of patients | 78.2 [73.3 to 82.5] | 82.7 [78.1 to 86.6]
Statistical Analysis 1: Comparison: Palonosetron and Placebo to Ondansetron vs Ondansetron and Placebo to Palonosetron; The null hypothesis (H0) was stated as: • H0 : CR 0-24 hr palonosetron - CR 0-24 hr ondansetron <-10% The alternative hypothesis (H1) was stated as: • H1 : CR 0-24 hr palonosetron - CR 0-24 hr ondansetron >-10% A power of 80% was used for sample size computation; Test type: Non-Inferiority or Equivalence — For the primary efficacy analysis, the confidence interval (CI) was built on the FAS using the stratum adjusted Mantel-Haenszel (MH) method with correction of continuity. The non-inferiority margin was -10%; Risk Difference (RD) = -4.4, 95% CI 2-sided [-10.5 to 1.7]

2. Secondary Outcome: Proportion of Patients With no Vomiting
Description: Time 0 (T0) was defined as the time when the patient wakes up and is able to show any active reaction postoperatively.
Time Frame: 0-24 hours after T0
Population: The Full Analysis Set (FAS) population.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Palonosetron and Placebo to Ondansetron | Ondansetron and Placebo to Palonosetron
Number analyzed (Participants) | 331 | 330
percentage of patients | 83.1 [78.5 to 86.9] | 87.6 [83.4 to 90.8]

3. Secondary Outcome: Proportion of Patients Without Emetic Episodes
Description: An emetic episode was defined as one or more continuous vomits (expulsion of stomach contents through the mouth) or retches (an attempt to vomit that is not productive of stomach contents). Time 0 (T0) was defined as the time when the patient wakes up and is able to show any active reaction postoperatively.
Time Frame: 0-24 hours after T0
Population: The Full Analysis Set (FAS) population.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Palonosetron and Placebo to Ondansetron | Ondansetron and Placebo to Palonosetron
Number analyzed (Participants) | 331 | 330
percentage of patients | 80.1 [75.3 to 84.1] | 83.9 [79.4 to 87.6]

4. Secondary Outcome: Proportion of Patients Without Antiemetic Rescue Medication
Description: Rescue medications are any medications with potential antiemetic effect taken in the 24 hours after patient wake-up from anaesthesia (T0).Time 0 (T0) was defined as the time when the patient wakes up and is able to show any active reaction postoperatively.
Time Frame: 0-24 hours after T0
Population: The Full Analysis Set (FAS) population.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Palonosetron and Placebo to Ondansetron | Ondansetron and Placebo to Palonosetron
Number analyzed (Participants) | 331 | 330
percentage of patients | 93.1 [89.6 to 95.4] | 96.4 [93.6 to 98.0]

5. Secondary Outcome: Proportion of Patients Without Nausea (Patient Aged > 6 Years)
Time Frame: 0-24 hours after T0
Population: The Full Analysis Set (FAS) population aged ≥ 6 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Palonosetron and Placebo to Ondansetron | Ondansetron and Placebo to Palonosetron
Number analyzed (Participants) | 185 | 183
percentage of patients | 83.2 [76.9 to 88.2] | 82.0 [75.5 to 87.1]

ADVERSE EVENTS:
Arm/Group | Palonosetron and Placebo to Ondansetron | Ondansetron and Placebo to Palonosetron
Serious Adverse Events (participants affected / at risk) | 4/331 | 11/330
Other Adverse Events (participants affected / at risk) | 234/331 | 225/330
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palonosetron and Placebo to Ondansetron (N=331) | Ondansetron and Placebo to Palonosetron (N=330)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 5 (6)
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Palatal oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Palonosetron and Placebo to Ondansetron (N=331) | Ondansetron and Placebo to Palonosetron (N=330)
Procedural pain (Injury, poisoning and procedural complications) | 147 (149) | 123 (126)
Pyrexia (General disorders) | 22 (22) | 25 (30)
Pain (General disorders) | 15 (16) | 15 (16)
Hyperthermia (General disorders) | 2 (2) | 12 (19)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 27 (28) | 37 (39)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Vomiting (Gastrointestinal disorders) | 5 (5) | 10 (12)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 8 (8)
Headache (Nervous system disorders) | 4 (4) | 10 (10)
Scar (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4)
Ear pain (Ear and labyrinth disorders) | 6 (6) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If Sponsor does not submit a publication regarding the study to a journal within 12 months from study data analysis completion, the Investigator may publish an analysis of the study data collected as a result of the conduct of the study by the Investigator. The Investigator shall ensure that at least 60 days prior to submitting/presenting a manuscript/material relating to study to publishers a copy of all manuscripts/materials is provided to the Sponsor to allow the Sponsor sixty days to review.